CLINICAL TRIAL: NCT02389998
Title: Evaluation of the Efficacy of Open Label Placebo in Children With FGIDs (Functional Gastrointestinal Disorders)
Brief Title: Efficacy of Open Label Placebo in Children With FGIDs
Acronym: Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Samuel Nurko, Attending Physician; Director, Center for Motility and Functional Gastrointestinal Disorders, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P00003158
Record Dates: First submitted 2015-02-25; First posted 2015-03-17 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Functional Abdominal Pain; Functional Dyspepsia; Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
Keywords: Functional Pain; Abdominal Pain; Irritable Bowel Syndrome; IBS; Functional Dyspepsia; FGID; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Abdominal Pain | interventions — Hyoscyamine

STUDY DESIGN:
Masking Description: Open placebo. No masking

ARMS (2):
- Placebo (Experimental): Arm 1: Subjects take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary for a period of three weeks. Subjects will also have access to hyoscyamine as a rescue medication.
  Interventions: Other: Placebo Suspension; Drug: Hyoscyamine
- No Treatment (Other): Arm 2: Subjects receive no treatment but have access to hyoscyamine as a rescue medication.
  Interventions: Drug: Hyoscyamine

INTERVENTIONS:
Other: Placebo Suspension — The study is divided into three phases: 1 one-week baseline assessment followed by 2 three-week study phases (phase A and phase B). Phase A will require subjects to take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary. In phase B subjects will not take the placebo. After 3 weeks in initial phase (either Phase A or B), subjects will switch to the alternate phase and continue the study for another 3 weeks. Hyoscyamine is available as a rescue medication during Phase A and Phase B. Half of the subjects will be randomized to begin with Phase A and half will be randomized to begin with Phase B.
  Arms: Placebo
Drug: Hyoscyamine — While not an intervention of interest to our study, patients will have hyoscyamine available as a rescue medication throughout the study. This can be taken on a PRN basis for breakthrough pain a maximum of 4x daily.

SUMMARY:
This study is aimed at investigating the efficacy of placebo for symptom relief in children with abdominal pain related functional gastrointestinal disorders.

DETAILED DESCRIPTION:
The purpose of this research study is to see if prescribing an open label placebo to children with functional gastrointestinal disorders will help improve symptoms and their overall quality of life. Open label means you/your child are aware you are taking liquid placebo drops and not an active medication. Symptoms associated with functional gastrointestinal disorders (FGIDs) of children and adolescents are commonly encountered symptoms in general pediatrics and pediatric gastroenterology. The FGIDs the investigators are studying include functional abdominal pain, irritable bowel syndrome, and functional dyspepsia. The liquid placebo drops contain no active medication.

Recent research studies have shown improvement in gastrointestinal symptoms after taking liquid placebo drops in both children and adults with FGIDs. A randomized research study for a medication used to treat children with FGIDs showed a very significant placebo effect, meaning patients receiving placebo also experienced improvement in their symptoms. Randomized refers to the fact that subjects were randomly selected to receive either the study medication or placebo. A recent adult study gave adult patients a placebo and told them it was a placebo, and these adults also had significant symptom improvement. The goal of this study is to further explore using open label (or non-deceptive) placebo use to treat children with FGIDs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to 21 years.
2. Diagnosis of functional abdominal pain, irritable bowel syndrome or functional dyspepsia made by a pediatric gastroenterologist according to Rome III Criteria.
3. Mean daily intensity of pain of 25 mm in the week prior to the initiation of the study, based on the Visual Analogue Scale
4. Children will not be excluded if they are adhering to any specific diet. Children will be asked to report any specific established diet prior to the study or dietary modifications that could have been made during the course of the study.
5. Normal laboratory tests including complete blood count, erythrocyte sedimentation rate, albumin, serum amylase, lipase, liver enzymes, urine analysis, stool examination for occult blood and ova and parasites one month prior the initiation of the study. Urinary culture will be obtained if the symptoms or urinalysis suggest the possibility of a urinary infection.
6. Normal lactose breath test or history of lack of resolution of symptoms on a lactose-free diet (2 weeks).
7. Patients receiving psychological treatment, hypnosis, biofeedback or guided imagery will not be excluded of the study if those were started at least one month prior to the initiation of the study and are not planned to be discontinued during the length of the trial. Patients will need to be prescribed hyoscyamine (clinically indicated) to be considered for this study, as the placebo will be in addition to their prescribed medication.

Exclusion Criteria:

1. Inclusion criteria not met.
2. Evidence of organic gastrointestinal disease, hepatic disorders, urinary or cardiac disease.
3. Children below the 5th percentile for weight or height.
4. Hemoccult positive stools.
5. Patients with diagnosis of Inflammatory Bowel Disease, hyperthyroidism, CHF, cardiac arrhythmias, prostatic hypertrophy, autonomic neuropathy, biliary tract disease, children with spastic paralysis or chronic lung disease (we will consult a pulmonologist concerning the inclusion of children with chronic lung disease).
6. Patients who are taking any of the following drugs: AbobotulinumtoxinA, Acetylcholinesterase Inhibitors (Central), Cannabinoids, OnabotulinumtoxinA, Potassium Chloride, Pramlintide, RimabotulinumtoxinB, Secretin. Patients receiving antidepressant or anticholinergic drugs will be excluded from the study. PPIs will be allowed as long as the patient had been on a stable dose for at least 12 weeks.
7. Patients planning to change their diet during the time of the study will be excluded. Children will be asked to report any specific established diet prior to the study or dietary modifications that could have been made during the course of the study.
8. Patients planning to start psychological treatment, hypnosis, biofeedback, or guided imagery during the course of the study or have started any of these within the month prior to consent.
9. The participant is pregnant or is planning to become pregnant throughout the course of the research study

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nurko, MD, MPH, Principal Investigator — Physician, Boston Children's Hospital; Miguel Saps, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nurko S, Saps M, Kossowsky J, Zion SR, Di Lorenzo C, Vaz K, Hawthorne K, Wu R, Ciciora S, Rosen JM, Kaptchuk TJ, Kelley JM. Effect of Open-label Placebo on Children and Adolescents With Functional Abdominal Pain or Irritable Bowel Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):349-356. doi: 10.1001/jamapediatrics.2021.5750. PMID 35099543

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cross over study
Groups:
- Placebo First Crossover to no Treatment After 3 Weeks: Arm 1: Subjects take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary for a period of three weeks. Subjects will also have access to hyoscyamine as a rescue medication.
  Placebo Suspension: The study is divided into three phases: 1 one-week baseline assessment followed by 2 three-week study phases (phase A and phase B). Phase A will require subjects to take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary. In phase B subjects will not take the placebo. After 3 weeks in initial phase (either Phase A or B), subjects will switch to the alternate phase and continue the study for another 3 weeks. Hyoscyamine is available as a rescue medication during Phase A and Phase B. Half of the subjects will be randomized to begin with Phase A and half will be randomized to begin with Phase B.
  Hyoscyamine: While not an intervention of interest to our study, patients will have hyoscyamine available as a rescue medication throughout the study. This can be taken on a PRN basis for breakthrough pain a maximum of 4x daily.
- No Treatment First Crossover to Placebo After 3 Weeks: Arm 2: Subjects receive no treatment but have access to hyoscyamine as a rescue medication.
  Hyoscyamine: While not an intervention of interest to our study, patients will have hyoscyamine available as a rescue medication throughout the study. This can be taken on a PRN basis for breakthrough pain a maximum of 4x daily.
Period: Overall Study
Arm/Group | Placebo First Crossover to no Treatment After 3 Weeks | No Treatment First Crossover to Placebo After 3 Weeks
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — car accident | 1 | 0

BASELINE CHARACTERISTICS:
Population: 30 patients were analyzed
Groups:
- Placebo First Followed by no Treatment: Arm 1: Subjects take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary for a period of three weeks. Subjects will also have access to hyoscyamine as a rescue medication.
  Placebo Suspension: The study is divided into three phases: 1 one-week baseline assessment followed by 2 three-week study phases (phase A and phase B). Phase A will require subjects to take 1/4 teaspoon placebo suspension 2 times a day (morning and night), and a third dose if necessary. In phase B subjects will not take the placebo. After 3 weeks in initial phase (either Phase A or B), subjects will switch to the alternate phase and continue the study for another 3 weeks. Hyoscyamine is available as a rescue medication during Phase A and Phase B. Half of the subjects will be randomized to begin with Phase A and half will be randomized to begin with Phase B.
  Hyoscyamine: While not an intervention of interest to our study, patients will have hyoscyamine available as a rescue medication throughout the study. This can be taken on a PRN basis for breakthrough pain a maximum of 4x daily.
- No Treatment First Followed by Placebo: Arm 2: Subjects receive no treatment but have access to hyoscyamine as a rescue medication.
  Hyoscyamine: While not an intervention of interest to our study, patients will have hyoscyamine available as a rescue medication throughout the study. This can be taken on a PRN basis for breakthrough pain a maximum of 4x daily.
- Total: Total of all reporting groups
Arm/Group | Placebo First Followed by no Treatment | No Treatment First Followed by Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Functional abdominal pain [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was Mean Daily Pain
Description: Change in mean pain score comparing both treatment arms to the baseline using the Visual analogue scale. (Scale 0-100mm)
  The scale reflects severity of the pain going from no pain (0) to maximum pain (100mm). Therefore the higher the number the more severe the pain is
Time Frame: It will be assessed at the end of the 3-week and 6-week treatment periods (at the end of each treatment arm prior to crossover to the next arm of treatment)
Population: A total of 30 patients completed the study. All of them received placebo or no treatment in a randomized crossover study. All measurements during placebo are combined. All measurements during no treatment are combined. Statistcal models were adjusted for order of treatment
Measure: Mean (Standard Deviation); unit: pain scale by VAS in mm
Arm/Group | Placebo | No Treatment
Number analyzed (Participants) | 30 | 30
pain scale by VAS in mm | 39.9 (18) | 45.14 (14.7)
Statistical Analysis 1: Comparison: Placebo vs No Treatment; Test type: Superiority; p < 0.03, ANCOVA

2. Secondary Outcome: Use of Rescue Medications
Description: The number of medications used as rescue during each one of the periods of the study were counted
Time Frame: 3 weeks of placebo vs 3 weeks of no treatment
Population: All patients
Measure: Mean (Standard Error); unit: pill count number
Groups:
- Placebo: Patients during the placebo periods
- No Treatment: Patients during the no treatment period
Arm/Group | Placebo | No Treatment
Number analyzed (Participants) | 30 | 30
pill count number | 2.0 (2.95) | 3.8 (5.05)
Statistical Analysis 1: Comparison: Placebo vs No Treatment; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Clinical Global Improvement
Description: Compared clinical global improvement during each phase of the study The following question was used: Overall, how do you feel your problem is? (better, same, or worse)." Patients were then divided in 2 groups: improved (if they answered better) vs not improved (if they answered same/worse)
Time Frame: Following 1-week baseline and 3-week and 6-week treatment periods
Population: A total of 30 patients completed the study. All of them received placebo or no treatment in a randomized crossover study. All measurements during placebo are combined. All measurements during no treatment are combined. Statistical models were adjusted for order of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | No Treatment
Number analyzed (Participants) | 30 | 30
Participants
  Improvement | 14 | 9
  No improvement | 16 | 21
Statistical Analysis 1: Comparison: Placebo vs No Treatment; Test type: Superiority; p = 0.3, McNemar

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT02389998/Prot_SAP_000.pdf